CLINICAL TRIAL: NCT07373275
Title: Investigating Lifestyle Medicine Interventions for Adolescent Headache Relief
Brief Title: Adolescent Lifestyle Medicine Headache Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Jennifer Dubail, MD, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: mainehealth
Record Dates: First submitted 2025-12-17; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Headache, Migraine
Keywords: Lifestyle Medicine; Adolescent; Implementation Science; headache; migraine
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: This is an Implementation Science study to assess the feasibility of using Lifestyle Medicine Group Medical Visits for adolescents with headache. We are using two groups with a step wedge design; both groups are getting the same intervention.
Masking Description: No one will be masked in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Lifestyle Medicine Intervention Arm (Experimental): All participants will receive the Lifestyle Medicine Group Medical Visit intervention, whether they are in group 1 or group 2.
  Interventions: Behavioral: Lifestyle Medicine Group Medical Visits

INTERVENTIONS:
Behavioral: Lifestyle Medicine Group Medical Visits — Participants will attend a virtual, one-hour weekly lifestyle medicine group session with their peers for 7 weeks. Each session will address one pillar of Lifestyle Medicine: restorative sleep, healthy eating, stress management, physical activity, avoiding risky substances, and positive social connection. During each session, study team members will provide a short presentation of key components of that lifestyle intervention and meet with participants in small groups to discuss goals related to that pillar (i.e. eat 2 more vegetables a day for five days). During the course of these 7 weeks, participants will also keep a virtual daily headache journal; a link to this journal will be sent through an automated text with a HIPPA-compliant REDCap database. This will be sent daily at 5 pm.

SUMMARY:
The goal of this pilot clinical trial is to assess the implementation of a 7-week Lifestyle Medicine intervention for adolescents with headache. The main question it aims to answer is:

Is it feasible to implement a Lifestyle Medicine curriculum for adolescents with headache and secondarily, does this intervention show any signal for improving headache symptoms?

Participants will be divided into two groups based on the order of their enrollment. After consent, they will be asked to complete 3 symptom surveys: PedMIDAS-6w, PHQ-A and GAD-7, in addition to a Lifestyle Survey. They will attend group medicine visits virtually, facilitated by the study team. Each week will address a different tenant of Lifestyle Medicine (such as eating or sleep) and participants will create a SMART goal to work on for the week. At the end of the seven weeks, they will repeat these symptom and lifestyle surveys. During the seven weeks, they will also keep a daily symptom diary, which will be texted to their phones through a HIPPA-compliant RedCAP database.

DETAILED DESCRIPTION:
Lifestyle Medicine is a medical specialty that emphasizes the use of group medical visits to teach and reinforce intensive, evidence-based lifestyle interventions to prevent, treat, and reverse chronic conditions such as headache. Lifestyle Medicine is built on six key pillars: restorative sleep, healthy eating, stress management, physical activity, avoiding risky substances, and positive social connection. Lifestyle modifications, including improved sleep, diet, and exercise are increasingly recommended as first-line approaches for the treatment and prevention of pediatric headache. However, these modifications are often difficult to implement consistently in adolescents due to the lack of structured, developmentally tailored programs that guide behavior change and provide ongoing support.

Study Intervention: Each group will participate in a Zoom meeting with 2-3 members of the research team for 60 minutes once a week for a 7-week program. The first week will be an introduction to the Lifestyle Medicine intervention, a conversation about confidentiality and ground rules for participation in group medical visits. Parents/guardians will be invited to participate in the introduction week if they wish. Participants will be sent a daily link to allow them to complete a headache diary to keep for the duration of the 7-week intervention. In weeks 2 through 7, the sessions will each be focused on one of the 6 lifestyle medicine pillars (restorative sleep, healthy eating, stress management, physical activity, avoiding risky substances, and positive social connection). The sessions will consist of a short presentation about the pillar and the importance of the pillar in reducing symptoms of headache. This presentation will be followed by a group discussion about how aspects of that pillar relate to the participant's experience of headache. For example, during the conversation about sleep, participants could be asked to reflect on their own sleep habits (e.g. what time they go to bed, do they fall asleep right away, is there a TV or phone in their room, do they get woken by text messages, how does fragmented sleep affect them the following day with particular emphasis on headache symptoms). At the end of each visit, each participant will make a Lifestyle Medicine SMART goal pertaining to that week's pillar. A SMART goal is a well-defined objective that is Specific, Measurable, Achievable, Realistic and Time-bound. This goal setting will be done in small breakout groups with study team members; during the session about substance use, goal setting will be done one-on-one. Participants will be asked to collect data during the following week on how successful they were in achieving their SMART goal. They will also be asked to keep a record of their headache symptoms in the headache diary. Study team members will record the goal setting in the electronic medical record (EPIC) and keep study notes about the sessions weekly through RedCAP, which include a feasibility checklist as well as narrative data re: the Proctor Model (Acceptability, Appropriateness, Costs, Feasibility, Fidelity, Penetration, Sustainability).

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old
* Frequent episodic migraine headaches with our without aura (>4 months)
* Patient at MaineHealth Pediatric Neurology or MaineHealth Pediatrics Portland
* Current High School Enrollment
* English Speaking

Exclusion Criteria:

* Age <14 year or >18 years
* Diagnosis of eating disorder or Autism Spectrum Disorder
* PHQ-A scores of 20 or higher
* Intractable/daily headache
* Headache secondary to specific medical or neurological conditions (e.g. brain tumor, infection, trauma)
* Increase in prophylactic headache medication 6 weeks prior to the onset of intervention

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Attendance | From enrollment to end of treatment at 3 months
  For this outcome, we will track how often participants attend the group meetings. There will be seven group meetings to attend, one per week. Attendance will be tracked at each meeting by group facilitators. We will calculate the overall percentage of attendance for each participant over the seven weeks and report the mean percentage. We anticipate >75% attendance to be successful.
Headache Diary Completion | From enrollment to end of treatment at 3 months
  For this outcome, we will track how often participants attend the group meetings. There will be seven group meetings to attend, one per week. Attendance will be tracked at each meeting by group facilitators. We will calculate the overall percentage of attendance for each participant over the seven weeks and report the mean percentage. We anticipate >75% attendance to be successful.

SECONDARY OUTCOMES:
Positive Lifestyle Changes | From enrollment to end of treatment at three months
  For this outcome, participants will be taking the survey Pediatric Lifestyle Medicine Assessment for Headache. This survey assesses nutrition and sleep. They will take this survey at their intake appointment and 7 weeks following the conclusion group medical visit sessions. For sleep, we anticipate measuring success through an increase in one hour or more of sleep nightly over the course of three surveys; we anticipate measuring nutrition through a decrease in skipped breakfasts by 25%.
Headache Symptoms | From enrollment through 3 months.
  For this outcome, participants will be filling out a daily headache diary, texted automatically through RedCAP. The first question asks if they had a headache in the last 24 hours, yes or no. To calculate the presence of headache in participants, we will [Anya? How do we get our number and what does the number mean?] A logistic mixed effects regression model will be used with a fixed effect for day and a random effect for participant to determine if the odds of headache decreases over time.
Headache Severity | From enrollment through 3 months.
  or this outcome, participants will be filling out a daily headache diary, texted automatically through RedCAP. If participants answer yes to headache presence in the first question, they will be asked a series of other questions. One question asks about headache severity, using a Likert scale. To analyze this, we will assign absence of headache as 0, and assess improvement in severity over time using a linear mixed effects model with a fixed effect for day and a random effect for participant.
Headache Symptom Reduction | From enrollment through 3 months.
  For this outcome, participants will be taking a commonly, clinically-used headache symptom survey, the Peds-MIDAS. The Peds-MIDAS will be adapted to be taken at 6 week intervals (Peds-MIDAS6w). Participants will take the Peds-MIDAS6w at their intake session, at their final group session, and 7 weeks following the completion of the study. They will score from 0-50, with 50 being the most severe. To assess improvement over time, we will use a linear mixed effects regression model with a random effect for participant, with success measured by a decrease in patient score by 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dubail, M.D., Principal Investigator — MaineHealth; Helis Jason, M.D., Principal Investigator — MaineHealth

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.